CLINICAL TRIAL: NCT06885788
Title: Comparative Study on the Effect of Uterine Round Ligament Preservation Vs Resection in Laparoscopic Inguinal Hernia Repair in Women： a Multicenter,Stratified Randomized Controlled Trial
Brief Title: Uterine Round Ligament Preservation Vs Resection in Laparoscopic Inguinal Hernia Repair in Women：A Multicenter,Stratified Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanchong Central Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025006
Record Dates: First submitted 2025-03-08; First posted 2025-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Inguinal Hernia; Laparoscopic Surgery; Randomized Controlled Trial
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Patients with unilateral hernia who did not give birth,the uterine round ligament resection group (Experimental): Both groups underwent laparoscopic inguinal hernia repair,the resection group removed the uterine round ligament.(Patients with unilateral hernia who did not give birth)
  Interventions: Procedure: To remove the uterine uterine ligament
- Patients with unilateral hernia who did not give birth,the uterine round ligament preservation group (No Intervention): Both groups underwent laparoscopic inguinal hernia repair,the preservation group retained the uterine round ligament.(Patients with unilateral hernia who did not give birth)
- Patients with unilateral hernia who have given birth,the uterine round ligament resection group (Experimental): Both groups underwent laparoscopic inguinal hernia repair,the resection group removed the uterine round ligament.(Patients with unilateral hernia who have given birth)
  Interventions: Procedure: To remove the uterine uterine ligament
- Patients with unilateral hernia who have given birth,the uterine round ligament preservation group (No Intervention): Both groups underwent laparoscopic inguinal hernia repair,the preservation group retained the uterine round ligament.(Patients with unilateral hernia who have given birth)
- Patients with bilateral hernias who have given birth,the uterine round ligament resection group (Experimental): Both groups underwent laparoscopic inguinal hernia repair,the resection group removed the uterine round ligament.(Patients with bilateral hernias who have given birth)
  Interventions: Procedure: To remove the uterine uterine ligament
- Patients with bilateral hernias who have given birth,the uterine round ligament preservation group (No Intervention): Both groups underwent laparoscopic inguinal hernia repair,the preservation group retained the uterine round ligament.(Patients with bilateral hernias who have given birth)
- Patients with bilateral hernia who did not give birth,the uterine round ligament resection group (Experimental): Both groups underwent laparoscopic inguinal hernia repair,the resection group removed the uterine round ligament.(Patients with bilateral hernia who did not give birth)
  Interventions: Procedure: To remove the uterine uterine ligament
- Patients with bilateral hernia who did not give birth,the uterine round ligament preservation group (No Intervention): Both groups underwent laparoscopic inguinal hernia repair,the preservation group retained the uterine round ligament.(Patients with bilateral hernia who did not give birth)

INTERVENTIONS:
Procedure: To remove the uterine uterine ligament — Both groups underwent laparoscopic inguinal hernia repair. The preservation group retained the uterine round ligament, while the resection group had it removed.
  Arms: Patients with bilateral hernia who did not give birth,the uterine round ligament resection group; Patients with bilateral hernias who have given birth,the uterine round ligament resection group; Patients with unilateral hernia who did not give birth,the uterine round ligament resection group; Patients with unilateral hernia who have given birth,the uterine round ligament resection group

SUMMARY:
This study aims to compare the clinical effects of uterine round ligament preservation versus resection in laparoscopic inguinal hernia repair in women.The primary outcomes included Time required for patient surgery.The secondary outcomes included Inguinal hernia recurrence,quality of life assessment,Indicators of postoperative recovery,, et al.

ELIGIBILITY:
Inclusion Criteria:

* ►Age : Female patients over 18 years of age without a childbearing requirement

  * Diagnosis and basis : Female patients diagnosed with Unilateral inguinal hernia.
  * agreed to participate in this study and signed the informed consent form.

Exclusion Criteria:

* ►Combined with severe heart, liver, kidney and other diseases.

  * pregnant or lactating women.
  * those with surgical contraindications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Time required for patient surgery | 20-120minutes
  Time required for patient surgery

SECONDARY OUTCOMES:
Inguinal hernia recurrence | 1 month, 3 months, 6 months,1year,2years,3years,6years
  the recurrence of inguinal hernia
Quality of life assessment | 3 months,6months,1year,2years,3years,6years
  Quality of life assessment:The international general quality of life scale (such as SF - 36, etc.) is used to evaluate the quality of life of patients at 3 months , 6months,1year,2years,3years and 6years after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanchong Central Hospital, Nanchong, Sichuan, China